CLINICAL TRIAL: NCT00722189
Title: Observational Study of the Efficacy, Safety and Tolerance of Travogen Cream (Isoconazole) and Travocort Cream (Isoconazole, Diflurcortolone) in the Treatment of Patients With Local Skin Mycosis of Various Etiology and Localization
Brief Title: Observational Study of Efficacy and Safety of Travogen Cream and Travocort Cream in the Treatment of Mycoses
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008/01850
Record Dates: First submitted 2008-07-14; First posted 2008-07-25 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2015-03

CONDITIONS: Skin Mycoses
Keywords: Mycoses
MeSH Terms: conditions — Dermatomycoses; Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: All patients treated

SUMMARY:
An assessment of the efficacy and safety of Travogen cream and Travocort cream in the treatment of local skin mycoses

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of skin mycosis

Exclusion Criteria:

* Allergies to study medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed skin mycoses
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of Travogen / Travocort in the treatment of skin mycoses / Travogen Cream and Travocort Cream will be prescribed by a physician | Baseline to end of study

SECONDARY OUTCOMES:
Patient satisfaction | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kashkin Clinical Research Mycological Institute, Saint Petersburg, Russia